CLINICAL TRIAL: NCT04650282
Title: A Phase II Randomized Controlled Double-Blind Clinical Trial of Sphenopalatine Ganglion (SPG) Block for Headache After Concussion
Brief Title: Sphenopalatine Ganglion Block for Headache After Concussion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Reassignment of PI to more intense clinical obligations prevents continuation of the trial.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Michael Popovich, Assistant Professor of Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00185200
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Concussion; Headache
Keywords: Concussions; headaches; sphenopalatine ganglion block
MeSH Terms: conditions — Brain Concussion; Headache | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Lidocaine in SphenoCath device (Experimental): One treatment will be given.
  Interventions: Combination Product: Lidocaine in SphenoCath device
- Saline Solution in SphenoCath device (Placebo Comparator): One treatment will be given.
  Interventions: Combination Product: Saline Solution in SphenoCath device

INTERVENTIONS:
Combination Product: Lidocaine in SphenoCath device — Participants will receive 2.5 cc of lidocaine 1% solution intranasally via a SphenoCath device into each nares.The portion of the procedure involving this device lasts approximately 30-60 seconds.
  Arms: Lidocaine in SphenoCath device
Combination Product: Saline Solution in SphenoCath device — Participants will receive saline solution via a SphenoCath device into each nares. The portion of the procedure involving this device lasts approximately 30-60 seconds.
  Arms: Saline Solution in SphenoCath device

SUMMARY:
This clinical trial will enroll participants to evaluate the effects of SPG block on post-traumatic headache. The study hypothesizes that patients that receive a SPG block with lidocaine vs. placebo (saline) will have a lower number of headache days in the week following the procedure, and will also report lower symptom scores.

Eligible participants will receive one treatment (SPG block) as well as complete surveys prior to and after receiving treatment (for a total of approximately 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a concussion and are greater than 14 days from the date of their injury.
* Experiencing greater or equal than 4 occurrences of headache per week lasting at least 1 hour per occurrence with a headache severity score greater or equal to 2 out of 6.

Exclusion Criteria:

* Allergy to local anesthetics of the amide type (for example (i.e.) lidocaine)
* Frequent epistaxis (i.e. more than one nose bleed per month),
* Bleeding disorders
* History of any of the following: nasal or facial fracture, nasal septal defect, any other craniofacial abnormality, hepatic disease, Adam-Stokes syndrome, Wolff-Parkinson-White syndrome, or severe degrees of sinoatrial, atrioventricular, or intraventricular heart block
* Pregnant
* Are at increased risk for methemoglobinemia (including patients with glucose-6-phosphate dehydrogenase deficiency, congenital or idiopathic methemoglobinemia, cardiac or pulmonary compromise, and concurrent exposure to oxidizing agents or their metabolites and drugs associated with methemoglobinemia)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Popovich, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request, I will share de-identified participant demographic information, outcome data, study protocol, statistical analysis plan, and informed consent form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be made available within 6 months of the study's conclusion, and will remain available for at least 5 years thereafter.
Access Criteria: Data will be made available if requested, pending a data use agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine in SphenoCath Device: One treatment was given.
  Lidocaine in SphenoCath device: Participants received 2.5 cc of lidocaine 1% solution intranasally via a SphenoCath device into each nares. The portion of the procedure involving this device lasted approximately 30-60 seconds.
- Saline Solution in SphenoCath Device: One treatment was given.
  Saline Solution in SphenoCath device: Participants received saline solution via a SphenoCath device into each nares. The portion of the procedure involving this device lasted approximately 30-60 seconds.
Period: Overall Study
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Customized [Count of Participants; unit: Participants]
  20 to 45 years of age | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Headache Severity Score
Description: Patients will rate their headache on a scale of 0 to 6, with 0 corresponding to "absent" and 6 corresponding to "severe."
Time Frame: 48 hours pre-SPG to 48 hours after SPG block
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: A rating scale of global improvement which participants use a seven-point scale ("1" = very much improved, "4" = no change, "7" very much worse). Participants will rate their change at two hours and 24 hours following the SPG block procedure.
Time Frame: 2, 24 hours after SPG block
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Change in the Number of Headache Occurrences
Description: The number of headache episodes over the one week prior to the SPG block compared to one week after the procedure.
Time Frame: 1 week before SPG block, up to 1 week post SPG block
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Headache Occurrences Within 48 Hours pre-and 48 Hours Post-SPG Block
Description: The number of headache episodes prior to the SPG block to after the procedure.
Time Frame: 48 hours pre SPG to 48 hours post block
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Headache Occurrences Within 1 Week Pre- and 1 Week Post-SPG Block
Description: The number of headache episodes over the one week prior to the SPG block to one week after the procedure.
Time Frame: 1 week before SPG block up to 1 week post SPG block
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mean Change in Headache Hours Per Day
Description: The number hours with headache 1 week prior to the SPG block and for up to 1 week after the procedure.
Time Frame: 1 week before SPG block, up to 1 week post SPG block
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mean Headache Hours Per Day Within 48 Hours Pre- and 48 Hours Post-SPG Block
Time Frame: 48 hours pre SPG up to 48 hours post SPG
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mean Headache Hours Per Day Within 1 Week Pre and 1 Week Post Block
Time Frame: 1 week before SPG block to 1 week post SPG block
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Mean Change in the Number of Days With Headache
Time Frame: 1 week before SPG block, up to 1 week post SPG
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Mean Number of Days With Headache in the1 Week Post-SPG Block Compared to 1 Week Pre-SPG Block.
Time Frame: 1 week before SPG block up to 1 week post SPG
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Mean Change in As-needed Headache Treatment Uses
Description: Patients will be asked to report the number of uses of as-needed headache medications used in the one week prior to the SPG block and after SPG block for up to one week after the procedure.
Time Frame: 1 week before SPG block to 1 week post SPG block
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Mean As-needed Headache Treatment Uses Within 48 Hours Pre- and 48 Hours Post-SPG
Description: as for outcome 11
Time Frame: 48 hours before SPG block to 48 hours post SPG block
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Mean As-needed Headache Treatment Uses Within 1 Week Pre and 1 Week Post Block
Description: as for outcome 11
Time Frame: 1 week before SPG block up to 1 week post SPG block
Population: Because only one participant was involved in each arm, showing data could violate privacy interests.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 Weeks: AE data was collected prior to and a week following procedure.
Arm/Group | Lidocaine in SphenoCath Device | Saline Solution in SphenoCath Device
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT04650282/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT04650282/ICF_001.pdf